CLINICAL TRIAL: NCT00504283
Title: An Analgesia Protocol for Acute Renal Colic in the DHMC Emergency Department
Brief Title: An Analgesia Protocol for Acute Renal Colic in the Emergency Department
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CPHS 20569
Record Dates: First submitted 2007-07-17; First posted 2007-07-19 (Estimated); Last update posted 2007-10-18 (Estimated); Status verified 2007-10

CONDITIONS: Kidney Stone
Keywords: Renal colic, pain, protocol, emergency department
MeSH Terms: conditions — Kidney Calculi; Renal Colic; Pain; Emergencies | interventions — Ketorolac Tromethamine; Morphine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Toradol
Drug: Morphine

SUMMARY:
An analgesia protocol for acute renal colic will lead to faster significant reductions in pain than prior practice.

DETAILED DESCRIPTION:
A retrospective study was performed that assessed the time to significant analgesia and medications used to achieve analgesia in the DHMC ED. Based upon this a prospective pain management protocol was designed and we will track the difference in time to significant pain relief between the two groups.

ELIGIBILITY:
Inclusion Criteria:

* Kidney stone on stone protocol CT scan
* Acute pain from a kidney stone

Exclusion Criteria:

* Age < 18 or > 65
* Pregnant women
* Contraindications to NSAID's or opiates

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2007-02; Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
Time to significant pain relief | Within emergency department

CONTACTS AND LOCATIONS:
Overall Officials: Peter L Steinberg, MD, Principal Investigator — DHMC dept of Urology
Locations (1):
- DHMC, Lebanon, New Hampshire, United States